CLINICAL TRIAL: NCT04353167
Title: Examination of the Relationship Between Foot - Body Posture and Balance and Gait in Duchenne Muscular Dystrophy
Status: Completed | Type: Observational
Sponsor: Hacettepe University (Other)
Responsible Party: Principal Investigator, Güllü AYDIN YAĞCIOĞLU, Principal Investigator, Hacettepe University
Other Study IDs: GO19548
Record Dates: First submitted 2020-04-16; First posted 2020-04-20 (Actual); Last update posted 2022-07-27 (Actual); Status verified 2022-07

CONDITIONS: Foot Posture; Balance; Gait Disorders, Neurologic; Body Posture
MeSH Terms: conditions — Gait Disorders, Neurologic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: observational evaluation — Patients will be evaluated only observationally without intervention

SUMMARY:
Foot and body postures of patients with DMD will be evaluated. Foot structure characteristics such as foot length, metatarsal width, calcaneal valgus angle will be calculated for the foot posture. Also, the Foot Posture Index (FPI-6) scale will be used. The body posture will be evaluated with the New York Posture Scale. Many gait characteristics such as step length, cadence, support surface of the patients will be determined with GaitRite instrumented walkway. Patients' balance assessment will be evaluated with Bertec Balance Advantage. The statistical analysis method will determine the relationship between foot and body posture and gait and balance.

ELIGIBILITY:
Inclusion Criteria:

1. To be between 5-13 years old
2. Being at level I or II according to Brooke Lower Extremity Functional Classification Scale
3. In the balance assessment, there should be at least 90 degrees of joint range of motion in the ankle to provide base contact on the force platform.
4. Agree to participate in the research voluntarily

Exclusion Criteria:

1. Having serious mental and psychological problems,
2. Failure to cooperate adequately with the physiotherapist making the evaluations,
3. Severe contracture in lower extremities,
4. Any injury and / or surgery of the lower extremities in the past 6 months.

Ages: 5 Years to 13 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Child
Study Population: Study population include just patients with Duchenne Muscular Dystrophy
Sampling Method: Non-Probability Sample
Enrollment: 38 (Actual)
Dates: Start 2020-03-15 (Actual); Primary Completion 2022-04-15 (Actual); Study Completion 2022-06-15 (Actual)

PRIMARY OUTCOMES:
Gait instrumented walkway (GaitRite) | 10 minutes
  The GAITRite® system mat was positioned on the floor and connected to a laptop computer, with a 2 m acceleration/deceleration walkway at either end. Subjects were asked to walk at their typical speed to the designated end of the walkway.
Bertec Balance System (Bertec) | 10 minutes
  The system consists of a 20 × 20-inch platform at ground level connected to a laptop computer. The balance plate detects body sway based on the pressure that the subject's feet apply to the plate surface. For testing, each subject stood for 10 seconds under 4 different testing conditions. The first two conditions were eyes open and eyes closed on the balance plate itself, defined as normal stability - eyes open (NSEO) and normal stability - eyes closed (NSEC). These were followed by the patient standing on a 4-inch thick foam rubber pad while on the balance plate. These were labeled as perturbed stability - eyes open (PSEO) and perturbed stability - eyes closed (PSEC). The primary measure assessed by the balance plate for each condition was maximum center of pressure excursion or COP (a distance measured in inches of the major axis of an ellipse calculated along the axis of maximum excursion).

SECONDARY OUTCOMES:
Foot Posture Index - 6 | 10 minutes
  The Foot Posture Index - 6 (FPI-6) was evaluated with each child standing and using the original protocol. FPI-6 values ranged from -2 to +2 for each of the six criteria and from -12 to +12 for the total score, indicative of position of each foot along the supinated to pronated continuum of foot posture.
NewYork Posture Scale | 10 minutes
  The assessment of posture was done by New York Posture Rating Scale in which subjects were asked to stand in position of comfort and look forward on the wall at their eye level in order to establish a level head position. Then the plumb line was kept slightly anterior to right malleolus for assessing posture in sagittal plane and at midpoint between the feet for assessing in the frontal plane. Scoring is done as 5, 3, 1 for no deviation, some deviation and marked deviation respectively for each 13 criteria in the rating scale of which components are head, shoulder, spine, hip, feet, arches in the frontal plane and head, chest, shoulder, upper back, trunk, abdomen and low back in the sagittal plane.

CONTACTS AND LOCATIONS:
Overall Officials: Güllü Aydın Yağcıoğlu, PhD, Principal Investigator — Hacettepe University
Locations (1):
- Hacettepe University, Ankara, Sıhhiye, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Aydin Yagcioglu G, Yilmaz O, Alemdaroglu Gurbuz I, Bulut N, Karaduman A, Ozkal O, Topuz S. Examination of the relationship between foot-body posture and balance and gait in Duchenne muscular dystrophy. Ir J Med Sci. 2023 Aug;192(4):1883-1888. doi: 10.1007/s11845-022-03178-5. Epub 2022 Oct 7. PMID 36205913